CLINICAL TRIAL: NCT03485079
Title: A Prospective, Multiple Center, Cohort Study of Prediction Model on Sudden Cardiac Death and Devices Development by Automatic Analysis From 24h Electrocardiogram in China
Brief Title: A Prospective,Multiple Center,Cohort Study of Prediction Model on Sudden Cardiac Death and Devices Development by Automatic Analysis From 24h Electrocardiogram in China
Acronym: PM-SCD CHINA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Jingfeng Wang (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Fudan University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor-Investigator, Jingfeng Wang, secretary of the party committee, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Other Study IDs: [2018]SYSEC-KY-KS-025
Record Dates: First submitted 2018-03-20; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, multicenter, cohort study. The study will be completed in three phases.

The first phase aims to establish SCD PW marker and PW score scoring system

1. Use big data processing techniques to find out the differences between survivors with ventricular arrhythmias and normal controls. Find out the SCD Pre-warning ECG Marker (PW marker).
2. Establish SCD Pre-warning risk score system according to traditional SCD risk factors, clinical characteristics of patients and abnormal electrocardiogram indicators.
3. According to the established SCD PW marker and PW score scoring system, the original group of patients are classified and scored. After five years of follow-up with sustained ventricular tachycardia or ventricular fibrillation as the primary end point and sudden cardiac death as the secondary endpoint, Kaplan-Meier are used to calculate the mortality rate of sudden cardiac death and Kaplan-Meier survival analysis. The COX proportional hazards regression model is used to further determine and evaluate the SCD predictive value of PW marker and PW score risk factor scoring system.

The second phase is to validate the established PW marker and PW score system models and evaluate the SCD predictive value of it. This stage is divided into two parts:

1. Patients enrolled in traditional high-risk ventricular arrhythmia, will be divided into PW marker positive group and PW marker negative group and join in a 5-year follow-up. Kaplan-Meier is used to calculate the mortality rate of sudden cardiac death and Kaplan-Meier survival analysis is performed to further verify the early warning effect of PW marker on SCD.
2. Patients will be divide into three groups including the low-risk group, middle-risk group and high-risk group according to the PW score risk factor scoring system and join in a 5-year follow-up. Kaplan-Meier is used to calculate the mortality rate of sudden cardiac death, and Kaplan-Meier survival analysis is used to further verify the early warning effect of PW score scoring system on SCD.

The third stage is the development stage of SCD early warning equipment. This stage will conduct clinical translational medical studies of PW marker and PW score based on the previous study and develop PW marker and PW score as portable SCD warning device and/or mobile phone APP which will be applied to the clinic for early warning diagnosis of SCD.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, cohort study. The study will be completed in three phases.

The first phase is a prospective, multi-center, cohort study of the SCD early warning model. This phase is divided into three parts:

1. Use big data processing techniques to find out the differences between survivors with ventricular arrhythmias and normal controls. Find out the SCD Pre-warning ECG Marker (PW marker), and determine the reasonable threshold of its early warning.
2. Establish SCD Pre-warning risk score system according to traditional SCD risk factors, clinical characteristics of patients and abnormal electrocardiogram indicators.
3. According to the established SCD PW marker and PW score scoring system, the original group of patients are classified and scored. After five years of follow-up with sustained ventricular tachycardia or ventricular fibrillation as the primary end point and sudden cardiac death as the secondary endpoint, Kaplan-Meier are used to calculate the mortality rate of sudden cardiac death and Kaplan-Meier survival analysis. The COX proportional hazards regression model is used to further determine and evaluate the SCD predictive value of PW marker and PW score risk factor scoring system.

The second phase is a prospective, multicenter, high-risk cohort study of SCD. It is used to validate the established PW marker and PW score system models and evaluate the SCD predictive value of it.

This stage is divided into two parts:

1. Patients enrolled in traditional high-risk ventricular arrhythmia, will be divided into PW marker positive group and PW marker negative group and join in a 5-year follow-up with sustained ventricular tachycardia or ventricular fibrillation as the primary end point and sudden cardiac death as the secondary endpoint. Kaplan-Meier is used to calculate the mortality rate of sudden cardiac death and Kaplan-Meier survival analysis is performed to further verify the early warning effect of PW marker on SCD.
2. Patients will be divide into three groups including the low-risk group, middle-risk group and high-risk group according to the PW score risk factor scoring system and join in a 5-year follow-up with sustained ventricular tachycardia or ventricular fibrillation as the primary end point and sudden cardiac death as the secondary endpoint. Kaplan-Meier is used to calculate the mortality rate of sudden cardiac death, and Kaplan-Meier survival analysis is used to further verify the early warning effect of PW score scoring system on SCD.

The third stage is the development stage of SCD early warning equipment. This stage will conduct clinical translational medical studies of PW marker and PW score based on the previous study and develop PW marker and PW score as portable SCD warning device and/or mobile phone APP which will be applied to the clinic for early warning diagnosis of SCD.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with recorded ventricular tachycardia, ventricular fibrillation or cardiac arrest meet one of the following conditions:

  1. survivors with cardiac arrest(including correct electrotherapy of ICD with ATP and electrical cardioversion)owing to non-reversible causes of ventricular fibrillation or hemodynamically unstable sustained ventricular tachycardia.
  2. Patients who suffer the underlying organic heart disease with spontaneous sustained ventricular tachycardia (including correct ICD therapy including ATP and cardioversion)

     1. more than 40 days after myocardial infarction , LVEF ≤ 0.35 with grade II or III cardiac function or more than 40 days after myocardial infarction, LVEF ≤ 0.30, with grade I cardiac function;
     2. non-ischemic cardiomyopathy, grade II or III heart function, LVEF ≤ 0.35;
     3. hereditary arrhythmia diseases: a group inherited diseases including long QT syndrome, short QT syndrome and Brugada syndrome, etc with arrhythmia, syncope and sudden death as the main clinical manifestations and cardiac gene mutation which encodes ion channels and their regulatory protein as the reason.

        long QT syndrome: electrocardiogram on the surface indicates QTc longer than 440 ms, accompanied by rapid ventricular arrhythmia, clinical symptoms of syncope and sudden death, without organic heart disease, except for acquired QT extension caused by electrolyte disorder and medication.

        short QT syndrome: electrocardiogram on the surface indicates QTc less than 300 ms, accompanied by rapid ventricular arrhythmia, clinical manifestations of syncope and sudden death, without organic heart disease, except for acquired etiology such as electrolyte disturbance and sympathetic stimulation.

        brugada syndrome: electrocardiogram on the surface suggests that the ST segment of leads V1-V3 is descending or saddle-shaped, accompanied by right bundle branch block, rapid ventricular arrhythmia, syncope, and sudden death without organic heart disease and ST-T changes due to other factors.

        catecholamine sensitive ventricular tachycardia: healthy individuals with no cardiac structural abnormalities and normal QTc suffer typical bidirectional, polymorphic ventricular tachycardia during exercise treadmill test or intravenous isoproterenol injection.
     4. hypertrophic cardiomyopathy: asymmetric ventricular septum hypertrophy> 15mm, or symmetrical hypertrophy ventricular septum thickness / left ventricular posterior wall thickness < 1.3 and left ventricular diastolic compliance decreased with or without left intraventricular or outflow obstruction confirmed by examination (including echocardiography, left ventricular angiography, cardiac MRI or cardiac CT, etc.).Heart changes caused by hypertension, aortic stenosis and other diseases need to be excluded.

Note: The above arrhythmia must be clearly recorded, including course records, nursing records, electrocardiogram, Holter, bedside ECG monitoring, telemetry ECG monitoring, portable ECG recorder, implanted device with program control data, including ECG Event recorders, pacemakers,ICDs, etc.

* 2.health checkers:physical examination patients without history of structural heart disease such as coronary heart disease or cardiomyopathy
* 3.patients or health checkers can learn to use microelectrocardiograph device after simple technical training;
* 4.patients or legal representatives or health checkers are willing and able to sign informed consent

Exclusion Criteria:

* 1.people who are pregnant or ready to become pregnant
* 2.people who are unable or unwilling to follow the study protocol and complete follow-up
* 3.people with uncontrolled hyperthyroidism and hypothyroidism, severe infection, severe hepatic and renal insufficiency (ALT≧3 times, or/and eGFR≦30mL/min calculated by any formula), malignancy, etc.
* 4.people with all kinds of idiopathic ventricular tachycardia diagnosed by electrocardiogram or electrophysiological examination, including idiopathic ventricular tachycardia in special parts such as left posterior branch, left anterior branch, right ventricular outflow tract, left ventricular outflow tract, etc.
* 5.people with various structural heart diseases, including various congenital heart diseases, rheumatic or senile heart valve disease
* 6.people with acute or subacute infective endocarditis, acute viral myocarditis
* 7.people with pulmonary arterial hypertension caused by right ventricular dysfunction alone, by UCG or right heart catheter examination PASP ≧ 40mmHg
* 8.people with severe electrolyte imbalance, acid-base imbalance
* 9.people with cardiac arrest caused by various severe bradyarrhythmias
* 10.people with known allergic reactions to adhesives or hydrogels
* 11.people whose skin cannot be pasted by electrode beacuse of a recent surgery.
* 12.people who are participating in other clinical trials and may affect the data collection of this study
* 13.people who have other situations that are not suitable for joining the group

Exit criteria:

* 1.people participating in the study can withdraw from the study at any time
* 2.people ask researchers for their desire to terminate the study
* 3.if the study jeopardizes the patient's health, the researcher can decide at any time to let the patient withdraw from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with recorded ventricular tachycardia, ventricular fibrillation or cardiac arrest and patients with traditional high-risk ventricular arrhythmia or health checkers in Sun Yat-sen Memorial Hospital, Sun Yat-sen University. Informed consent must be obtained for all of the included people.
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2018-04-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
SCD Pre-warning ECG Marker (PW marker) | baseline
  Use big data processing techniques to find out the differences between survivors with ventricular arrhythmias and normal controls
rate of sustained ventricular tachycardia or ventricular fibrillation | baseline and 5 years later
  Five years of follow-up with sustained ventricular tachycardia or ventricular fibrillation as the primary end point
rate of sudden cardiac death | baseline and 5 years later
  Five years of follow-up with sudden cardiac death as the secondary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Jingfeng Wang, M.D.,Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China